CLINICAL TRIAL: NCT06463457
Title: Comeback From Long coursE ADT With RElugolix and Darolutamide in Hormone-sensitive Prostate Cancer (CLEARED)
Brief Title: Comeback From Long coursE Androgen Deprivation Therapy (ADT) With RElugolix and Darolutamide (CLEARED)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Atish Choudhury, MD (Other)
Collaborators: Bayer (Industry); Pfizer (Industry); National Comprehensive Cancer Network (Network); Sumitomo Pharmaceuticals America (Industry)
Responsible Party: Sponsor-Investigator, Atish Choudhury, MD, Sponsor Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-217
Record Dates: First submitted 2024-06-11; First posted 2024-06-17 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Prostate Cancer; Advanced Prostate Cancer; Hormone Sensitive Prostate Cancer
Keywords: Hormone-Sensitive Prostate Cancer; Prostate Cancer; Advanced Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — darolutamide; relugolix

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Cohort 1 Short Pharmacokinetics (PK) (Experimental): Enrolled participants will complete study procedures as follows:
  * Cycle 1:
    * Day 1 of 28 Day Cycle: Predetermined dose of Relugolix 1x daily. First dose will be administered in-clinic.
    * Day 1 of 28 Day Cycle: Predetermined dose of Darolutamide 2x daily. First dose will be administered in-clinic.
  * Cycle 2 through End of Treatment:
    * Predetermined dose of Relugolix 1x daily.
    * Predetermined dose of Darolutamide 2x daily.
  * End of Treatment visit.
  * Follow Up: every 3 months for 18 months.
  Interventions: Drug: Darolutamide; Drug: Relugolix
- Cohort 2 Long Pharmacokinetics (PK) (Experimental): Enrolled participants will complete study procedures as follows:
  * Cycle 1:
    * Days 1, 2, 8 of 28 Day Cycle: Predetermined dose of Relugolix 1x daily. First dose will be administered in-clinic.
    * Days 1, 2, 8 of 28 Day Cycle: Predetermined dose of Darolutamide 2x daily. First dose will be administered in-clinic.
  * Cycle 2:
    * Day 1 of 28 Day Cycle: Predetermined dose of Relugolix 1x daily. First dose will be administered in-clinic.
    * Day 1 of 28 Day Cycle: Predetermined dose of Darolutamide 2x daily. First dose will be administered in-clinic.
  * Cycle 3 through End of Treatment:
    * Predetermined dose of Relugolix 1x daily.
    * Predetermined dose of Darolutamide 2x daily.
  * End of Treatment visit.
  * Follow Up: every 3 months for 18 months.
  Interventions: Drug: Darolutamide; Drug: Relugolix

INTERVENTIONS:
Drug: Darolutamide — Androgen receptor antagonist, tablet taken orally per protocol.
  Other Names: ODM-201; Bay 1841788; C19H19CIN6O2
Drug: Relugolix — Gonadotropin-releasing hormone (GnRH) receptor antagonist, tablet taken orally per protocol.
  Other Names: Orgovyx; RVT-601; TAK-385; 1-[4-[1-[(2,6-difluorophenyl)methyl]-5-[(dimethylamino)methyl]-3-(6-methoxypyridazin-3-yl)-2,4-dioxothieno[2,3-d]pyrimidin-6-yl]phenyl]-3-methoxyurea; C29H27F2N7O5S

SUMMARY:
This research study is being done to determine the rate of testosterone recovery after completing two years of treatment with the combination of relugolix and darolutamide as well as to assess the safety of the drugs when administered in combination.

The names of the drugs in this study are:

* Relugolix (a type of gonadotropin-releasing hormone receptor antagonist)
* Darolutamide (a type of androgen receptor antagonist)

DETAILED DESCRIPTION:
The aim of this single-arm phase 2 study is to assess testosterone recovery after completion of two years of combination treatment with relugolix and darolutamide and to describe safety, tolerability and pharmacokinetics of relugolix and darolutamide when administered in combination. Participants will select enrollment into one of two groups (Group 1 or Group 2). The purpose of Group 1 is to determine the amount of each drug in the bloodstream after 2 hours, 4 hours, and 8 hours of treatment, whereas the purpose of Group 2 is to determine the amount of each drug in the bloodstream after 1 day, 7 days, and 28 days of treatment.

The US Food and Drug Administration (FDA) has approved relugolix for the treatment of advanced prostate cancer.

The FDA has approved the combination of darolutamide with docetaxel for initial treatment of metastatic prostate cancer, that is, cancer that has spread to other parts of the body. The FDA has also approved darolutamide alone for treatment of non-metastatic castration-resistant prostate cancer, that is, cancer that has become resistant to testosterone lowering medications without evidence of spread of the cancer to other parts of the body that can be detected on Computerized Tomography (CT) or bone scans.

While darolutamide and relugolix can be prescribed together based on the FDA-approved indications of the individual drugs, this combination has not been approved by the FDA or formally tested in clinical trials.

The research study procedures include screening for eligibility, study treatment visits, questionnaires, and blood tests. Electrocardiograms (EKGs) will be performed if felt to be clinically indicated by the treating physician. Imaging using a Computerized Tomography (CT) scan, Magnetic Resonance Imaging (MRI) scan, bone scan, and/or Prostate-Specific Membrane Antigen Positron Emission Tomography (PSMA-PET) scan is required before starting study treatment, and will be performed after starting study treatment when felt to be clinically indicated by the treating physician.

Participants will receive study treatment of relugolix and darolutamide for 2 years and will be followed for 18 months after the treatment period.

It is expected that about 33 participants will take part in this research study.

Bayer AG, Pfizer, and Sumitomo Pharma America (SMPA), Inc. are funding this research study. Bayer and SMPA are providing the study drugs darolutamide and relugolix, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically or cytologically confirmed prostate cancer.
* Hormone-sensitive prostate cancer (with detectable prostate-specific antigen [PSA] > 0.02 ng/ml, testosterone ≥ lower limit of normal [LLN] per institutional assay) planned for two years of intensified androgen deprivation therapy per investigator discretion. This includes the following indications:

  * Treatment-naïve high risk lymph node-negative (N0) disease planned for primary radiation therapy
  * Treatment-naïve clinically pelvic lymph node positive (cN+) disease planned for primary radiation therapy
  * Pathologically pelvic lymph node positive (pN+) disease after prostatectomy planned for salvage radiation therapy
  * Regional nodal recurrence after prior local therapy (often in the context of radiation to lymph nodes)
  * Synchronous or metachronous low volume metastatic hormone sensitive prostate cancer (mHSPC) by Chemohormonal Therapy Versus Androgen Ablation Randomized Trial for Extensive Disease (CHAARTED) criteria planned for treatment interruption after 2 years (often in the context of radiation to sites of disease).
  * N.B: While CHAARTED criteria were established based on conventional imaging, patients who had PSMA PET imaging that would meet criteria for high volume disease (visceral metastases or ≥ 4 definitive bone metastases with at least one outside the axial skeleton) are excluded from this study.
* Prior hormonal therapy is permitted in the context of neoadjuvant/concurrent/adjuvant treatment with prior local therapy or biochemical recurrence by conventional imaging (for patients enrolling for recurrent rather than treatment-naïve disease), but patients must have had testosterone recovery to ≥ LLN at time of enrollment to this trial.
* Age ≥18 years. Children under 18 are excluded from this study as prostate cancer is a disease of adults.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤1 (Karnofsky ≥70%).
* Participants must meet the following organ and marrow function as defined below:

  * leukocytes ≥2500/mcL
  * absolute neutrophil count ≥1000/mcL
  * platelets ≥100,000/mcL
  * total bilirubin ≤ 1.5 institutional upper limit of normal (ULN) unless known or suspected Gilbert syndrome
  * aspartate aminotransferase (AST)/alanine aminotransferase (ALT) ≤2.5 × institutional ULN
  * glomerular filtration rate (GFR) ≥30 mL/min/1.73 m2 (based on Cockcroft-Gault formula, Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) refit formula, OR creatinine clearance based on 24 hour urine collection)
* Human immunodeficiency virus (HIV)-infected participants on effective anti-retroviral therapy (with no known or predicted drug-drug interactions with darolutamide and/or relugolix) with undetectable viral load within 6 months are eligible for this trial.
* For participants with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable. If suppressive therapy is indicated, there must be no known or predicted drug-drug interactions with darolutamide and/or relugolix.
* Participants with a history of hepatitis C virus (HCV) infection must have been treated and cured. For participants with HCV infection who are currently on treatment, they are eligible if there are no known or predicted drug-drug interactions with darolutamide and/or relugolix and they have an undetectable HCV viral load.
* Participants with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, participants should be class 2B or better.
* Ability to swallow oral medications.
* The effects of darolutamide and/or relugolix on the developing human fetus are unknown. For this reason and because oral hormonal agents are known to be teratogenic, participants must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while her partner is participating in this study, she should inform her treating physician immediately. Participants treated or enrolled on this protocol must also not donate semen or sperm and agree to use adequate contraception prior to the study, for the duration of study participation, and 3 months after completion of darolutamide and relugolix administration.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Participants who received prior systemic therapy for the disease state (high risk localized, lymph node positive, or low volume mHSPC) for which they are enrolling on this trial. Prior hormonal therapy is permitted for patients with recurrent disease after prior therapy.
* Participants who previously experienced any rise in PSA with castrate level testosterone (< 50 ng/dl).
* Participants who are receiving any other investigational agents for this condition.
* Participants with brain metastases, leptomeningeal disease, or metastases involving other visceral organs since these patients would be considered to have "high volume" metastatic disease by CHAARTED criteria.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to relugolix or darolutamide.
* Participants with predicted significant drug-drug interaction with darolutamide and/or relugolix are ineligible or must be monitored carefully as detailed below:

  * Participants receiving combined P-glycoprotein (P-gp) and strong CYP3A inducers (e.g. apalutamide, carbamazepine, fosphenytoin, phenobarbital, phenytoin, primidone, rifampin, rifapentine, and St. John's wort) or combined P-gp and moderate CYP3A4 inducers (e.g. efavirenz, rifabutin) are ineligible.
  * Participants receiving combined P-gp and strong CYP3A4 inhibitors (e.g. ketoconazole, itraconazole, posaconazole, clarithromycin, cobicistat, cyclosporine, tacrolimus, nelfinavir, ritonavir, lopinavir, saquinivir, tipranavir) are ineligible to enroll.
  * Participants receiving Breast cancer resistance protein (BCRP) substrates (e.g. glyburide, cimetidine, nitrofurantoin, dipyridamole, sulfasalazine, and rosuvastatin) are not excluded but participants should be monitored more frequently for adverse reactions to the BCRP substrate drug, and dose reduction of the BCRP substrate drug should be considered.
  * Participants receiving P-gp inhibitors are not excluded but participants must be able to dose the P-gp inhibitor at least 6 hours after relugolix dose during the conduct of the study. Participants unable to dose the P-gp inhibitor at least 6 hours after relugolix dose, or requiring twice daily or more frequent dosing of a P-gp inhibitor are ineligible.
  * Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated medical reference. As part of the enrollment/informed consent procedures, the participant will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the participant is considering a new over-the-counter medicine or herbal product.
* Participants with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia.
* Participants with psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant and nursing women are excluded from this study because they do not develop prostate cancer.
* Concurrent active malignancy. Patients with non-melanomatous skin cancer, superficial bladder cancer, cancer not needing active systemic therapy for at least 2 years and would not affect imaging assessments for prostate cancer, cancer for which the treating investigator deems the subject to be in remission, or any prior malignancy that was treated with curative intent (no evidence of disease for at least 3 years) are also permitted to enroll.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2024-12-13 (Actual); Primary Completion 2028-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
18-month Rate of Testosterone Recovery | 42 months (18 months after completion of 2 years of treatment)
  Rate of testosterone recovery (TR) defined as the proportion of participants achieving testosterone ≥ lower limit of normal by 18 months after completion of study treatment. Participants who withdrew from trial therapy (due to early progression, toxicity, patient/physician decision or death) before completing 2 years of treatment will be excluded from the analysis. Participants who require resumption of androgen deprivation, withdraw, are lost to follow-up, or die before 18 months of post-treatment follow up has been completed without having achieved testosterone recovery ≥ lower limit of normal beforehand will be included in the analysis and will be considered to be non-recovered.
Grade 3-5 Treatment-related Toxicity Rate | 24 months. AE collected on day 1 of each cycle (up to 26 cycles in total, each cycle is 28 days)
  All grade 3-5 adverse events (AE) with treatment attribution of possibly, probably or definitely related to study treatment based on Common Terminology Criteria for Adverse Events (CTCAE) version 5 are counted. Rate is the proportion of treated participants experiencing at least one of these adverse events as defined during the time of observation.

SECONDARY OUTCOMES:
Geometric Mean Ratio of Single-dose Cmax (highest concentration of drug) and Steady-state Ctrough (the concentration of drug in the blood immediately before the next dose is administered) | 29 days. Pharmacokinetic (PK) collection prior to the first dose of both drugs and then after 2 hours, 4 hours and 8 hours (Cohort 1) or after 24 hours, 7 days, and 28 days (Cohort 2) of uninterrupted dosing during cycle 1 (each cycle is 28 days).
  Geometric mean ratio (GMR) of single-dose Cmax (Cohort 1) and steady-state Ctrough (Cohort 2) of darolutamide and relugolix calculated as the geometric mean when administered in combination with the other agent divided by geometric mean when administered as monotherapy (historical control).
Rate of Treatment Discontinuation | 24 months. Treatment planned on day 1 of each cycle (up to 26 cycles in total, each cycle is 28 days)
  Rate of treatment discontinuation defined as the proportion of participants who discontinued treatment due to 1) adverse events, 2) disease progression, and 3) participant withdrawal.
Mean Functional Assessment of Cancer Therapy - Prostate (FACT-P) Score | 42 months. Collected at Cycle 1 day 1 (each cycle is 28 days), end of treatment (24 months), and end of study at 18 months after completion of treatment (42 months)
  The FACT-P is a well-established, 39-item questionnaire that was developed and validated specifically in participants with advanced prostate cancer. The FACT-P total score ranges from 0 to 156. Higher values of the FACT-P total and all subscales indicate a higher quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Atish Choudhury, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: atish_choudhury@dfci.harvard.edu. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu